CLINICAL TRIAL: NCT05014516
Title: Lung Structure-Function In SurVivors of Mild and SEvere COVID-19 Infection: 129Xe MRI For Rapid Evaluation and NExt-wave Healthcare Planning
Brief Title: Lung Structure-Function In SurVivors of Mild and SEvere COVID-19 Infection: 129Xe MRI
Acronym: LivCovidFree
Status: Terminated | Type: Observational
Why Stopped: Recruitment Challenges
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Western University (Other)
Responsible Party: Principal Investigator, Giles Santyr, Senior Scientist, The Hospital for Sick Children
Other Study IDs: 1000074027
Record Dates: First submitted 2021-07-30; First posted 2021-08-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: COVID-19 Respiratory Infection
Keywords: Lung MRI; 129Xenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm: Those participants who have experienced a documented case (documented by positive COVID19 test and/or clinical history) mild or severe COVID19 infection including those with symptoms and those who were hospitalized with COVID19 infection, all of whom are within 3 months post recovery
  Interventions: Drug: 129Xenon gas

INTERVENTIONS:
Drug: 129Xenon gas — Observational
  Other Names: Hyperpolarized tracer gas

SUMMARY:
In this study the Investigators aim to deploy UTE and HP 129Xe MRI for structural and functional evaluation of persistent lung abnormalities in COVID-19 survivors.

DETAILED DESCRIPTION:
What is COVID-19? The ongoing Coronavirus Disease 2019 (COVID-19) pandemic is caused when an individual is infected with the SARS-CoV-2 virus. This infection can result in pneumonia involving the small airways and alveoli (the tiny air sacs at the end of the airways that help oxygen get into the blood). COVID-19 can cause damage to the lungs, making it hard to breathe without medical help. To understand what is happening to a patient's lungs, doctors may use imaging tests such as chest x-rays or CT Scans (computed tomography). However, these types of tests may not tell the Investigators the whole story.

What is the purpose of the study? Led by The Hospital for Sick Children (SickKids), this study is being done to determine if MRI (magnetic resonance imaging) scans can tell the Investigators more about the lungs of people who had COVID-19. The Investigators will use a special type of MRI where participants breathe in a special gas (hyperpolarized xenon-129) before they have the MRI. This gas will help the Investigators to see' the lungs. The advantage of MRI scans is that there is no radiation involved in these types of images.

What is involved? In this study, participants will have an MRI of their lungs. The Investigators will examine these MRI scans to see if the Investigators can identify any changes in the structure or the function of the lung. If the Investigators do find any changes, they will see how these changes relate to other tests that have been conducted or other parts of the clinical story.

The participants will be asked to come to SickKids for 3 study visits. A fourth visit will be conducted via telephone. These visits will span over 3 years. Each study visit will take about 4 hours. If the participant is unable to attend one of the in-person visits, they will be given the option for a phone/virtual visit instead.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* Aged 12-70 years old
* Meets MRI screening criteria
* Diagnosed with COVID19, documented by positive COVID19 test (Nasopharyngeal swab or saliva swab) and are within 3 months post recovery*.

  * Recovery from COVID19 is defined as asymptomatic for at least 2 weeks prior to study visit 1 and screen negative based on SickKids guidelines.

Exclusion Criteria:

* Pregnant or lactating*
* A cold or flu within the last 2 weeks

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 40 participants age ≥ 12 and ≤70 years who experienced a documented case (documented by positive COVID19 test and/or clinical history) mild or severe COVID19 infection including those with symptoms and those who were hospitalized with COVID19 infection, all of whom are within 3 months post recovery.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Primary | 4 years
  Determine if 129Xenon MRI can detect abnormalities in COVID19 survivors 3 months, 6 months, 1 year and 2 years post infection.

SECONDARY OUTCOMES:
Secondary 2A (i) | 3.5 years
  Pulmonary function test: Spirometry to measure FEV1 (L)
Secondary 2A (ii) | 3.5 years
  Pulmonary function test: Plethysmography/Lung volumes to measure TLC (L)
Secondary 2A (iii) | 3.5 years
  Pulmonary function test: Diffusing Capacity Of The Lungs For Carbon Monoxide to measure DLCO
Secondary 2B | 3.5years
  6 minute walk test - The object of this test is to walk as FAR AS POSSIBLE for 6 minutes.
Secondary 2C | 3.5 years
  St. George's Respiratory Questionnaire: Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways
Secondary 2D | 3.5 years
  Dyspnea Score: it allows the patients to indicate the extent to which their breathlessness affects their mobility. The 1-5 stage scale is used alongside the questionnaire to establish clinical grades of breathlessness.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kooner HK, Wyszkiewicz PV, Matheson AM, McIntosh MJ, Abdelrazek M, Dhaliwal I, Nicholson JM, Kirby M, Svenningsen S, Parraga G. Chest CT Airway and Vascular Measurements in Females with COPD or Long-COVID. COPD. 2024 Dec;21(1):2394129. doi: 10.1080/15412555.2024.2394129. Epub 2024 Sep 2. PMID 39221567
- [Derived] Kooner HK, McIntosh MJ, Matheson AM, Abdelrazek M, Albert MS, Dhaliwal I, Kirby M, Ouriadov A, Santyr GE, Venegas C, Radadia N, Svenningsen S, Nicholson JM, Parraga G. Postacute COVID-19 Syndrome: 129Xe MRI Ventilation Defects and Respiratory Outcomes 1 Year Later. Radiology. 2023 Apr;307(2):e222557. doi: 10.1148/radiol.222557. Epub 2023 Feb 7. PMID 36749209
- [Derived] Kooner HK, McIntosh MJ, Matheson AM, Venegas C, Radadia N, Ho T, Haider EA, Konyer NB, Santyr GE, Albert MS, Ouriadov A, Abdelrazek M, Kirby M, Dhaliwal I, Nicholson JM, Nair P, Svenningsen S, Parraga G. 129Xe MRI ventilation defects in ever-hospitalised and never-hospitalised people with post-acute COVID-19 syndrome. BMJ Open Respir Res. 2022 May;9(1):e001235. doi: 10.1136/bmjresp-2022-001235. PMID 35584850